CLINICAL TRIAL: NCT04348396
Title: ReportAge-COVID Project: Clinical and Biological Predictors of COVID-19 Disease in Older Patients
Brief Title: Clinical and Biological Predictors of COVID-19 Disease in Older Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_01_2020
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: COVID-19; older people; SARS-CoV-2; frailty; physical function; biomarkers of inflammation
MeSH Terms: conditions — COVID-19; Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The surplus of serum and plasma in the blood samples taken from patients for routine examinations during hospitalization will be stored at -80°C at the BioGer biobank of IRCCS INRCA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients affected by COVID-19: The group taken into consideration consists of elderly patients hospitalized with diagnosed COVID-19.

SUMMARY:
The project is an observational, prospective study. Its aim is to deepen our understanding of COVID-19 in older patients hospitalized and diagnosed with COVID-19.

In particular, socioeconomic, diagnostic, biological, functional, therapy data will be collected at the patients' admission, during hospital stay, at the discharge and 1, 3, 6, 12 months after discharge.

Results and findings will help support changes in clinical practice and decision making, with the aim to reduce the use of healthcare services and the healthcare expenditure.

DETAILED DESCRIPTION:
Current knowledge about clinical and biological characteristics of COVID 19 among older people is very limited. A better comprehension of the clinical picture of older patients affected by COVID-19, (e.g. frailty, multimorbidity and polypharmacy patterns and functional performance) may significantly contribute to deepen our understanding of the clinical epidemiology knowledge of COVID-19 among hospitalized older people.

Therefore, the ReportAge-COVID project aims to collect - using a minimum clinical and biological data set - a series of data and indicators on the conditions of elderly patients that are suspected of having a compatible clinical picture or were confirmed positive for COVID-19. Data will be collected at the patients' admission, during hospital stay, at discharge and 1, 3, 6, 12 months after discharge.

In particular, the following specific pieces of information will be gathered:

* routinely collected demographic, socioeconomic, clinical, biological and diagnostic data
* frailty condition (by using the clinical frailty scale)
* assessment of the functional capacities through ADL and IADL tests
* health conditions; nutritional status; medications; treatments and procedures
* biomarkers of aging including cytokines and anti-inflammatory molecules, previously identified in a focus group of experts

Results and findings will help support changes in clinical practice and decision making, with the aim of reducing adverse outcomes, the worsening of health conditions in the elderly population, the use of healthcare services and, as a consequence, lower healthcare expenditure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COVID-19

Exclusion Criteria:

* no informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients 65 years old and above hospitalized for COVID-19
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive-epidemiological analysis of health conditions | Patients will be followed for the duration of hospital stay, an expected average of 20 days
  Collection of a set of data and indicators of the health conditions including personal data, clinical care, biological and diagnostic data, treatments/procedures and drug therapy

SECONDARY OUTCOMES:
Evaluation of frailty condition | At admission, at discharge, an expected average of 6 weeks and at 1, 3, 6, 12 months after discharge
  Clinical Frailty Scale (CFS). The CFS divides patients into 9 classes from very fit (CFS=1) to terminally ill (CFS=9)
Identification of biomarkers of inflammation | At admission, at discharge, an expected average of 6 weeks and at 1, 3, 6, 12 months after discharge
  Analysis for IL6, IL-10, IL-2, IL-7, Alpha 1 Antitrypsin, IP10, MCP1, MIP1 alpha, TNF alpha, IFN alfa, IFN beta
Assessment of functional capacity | At admission, at discharge, an expected average of 6 weeks and at 1, 3, 6, 12 months after discharge
  Activity of Daily Living (ADL). A summary score ranges from 0 (low function, dependent) to 6 (high function, independent)
Assessment of functional capacity | At admission, at discharge, an expected average of 6 weeks and at 1, 3, 6, 12 months after discharge
  Activity of Instrumental of Daily Living (IADL). A summary score ranges from 0 (low function, dependent) to 8 (high function, independent)
Evaluation of drug consumption | At admission, at discharge, an expected average of 6 weeks and at 1, 3, 6, 12 months after discharge
  Drugs prior to admission, drugs administered during hospital stay, prescribed drugs at discharge
Evaluation of inflamma-miRs | At admission, at discharge, an expected average of 6 weeks and at 1, 3, 6, 12 months after discharge
  Determination of miR-21, miR-146a, miR-155

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS INRCA Hospital, Ancona
  - IRCCS INRCA Hospital, Casatenovo
  - IRCCS INRCA Hospital, Fermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IRCCS INRCA website — http://www.inrca.it